CLINICAL TRIAL: NCT04396132
Title: The Effect of Head Tilt and Soft Surface on Virtual SVV in Normal Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Chief of Department, Pamukkale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4
Record Dates: First submitted 2020-05-17; First posted 2020-05-20 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Vestibular Nerve Diseases
MeSH Terms: conditions — Vestibulocochlear Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual SVV (Experimental): The subjects will be tested by virtual SVV. The deviation angle will be measured at 15, 30 and 45-degree head tilt to the left and right side while they are standing
  Interventions: Diagnostic Test: Subjective Visual Vertical with Virtual SVV instrument

INTERVENTIONS:
Diagnostic Test: Subjective Visual Vertical with Virtual SVV instrument — The deviation angle will be measured with 15, 30 and 45-degree head tilt to the left and right side while they are standing

SUMMARY:
The sense of gravity is one of the important input of our balance system. The utricle is the key structure on this subject but the contribution of the proprioceptive receptors is also important. The aim of this study is to measure the effect of different angles of head tilt and soft surface on SVV in healthy subjects with a new automated system.

DETAILED DESCRIPTION:
Two different settings will be used. In the first experiment, healthy subjects will make 15, 30, and 45-degree head tilt to the left and right side while they are standing. In every position, 3 measurements will be done. In the second experiment, 40 health subjects will make the same head maneuvers on the 20 cm thick soft surface. We will compare the effects of both head tilt and soft surface. All measurements will be done with a virtual SVV system(Interacoustics).

ELIGIBILITY:
Inclusion Criteria:

* No ear disease
* No neurologic disease
* No surgery for ear, brain or musculoskeletal system

Exclusion Criteria:

* Diabetes mellitus
* Drug use effective on central nervous system

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Subjective Visual Vertical | 1 month
  The measurement of deviation angle with 15, 30 and 45-degree head tilt to the left and right side while they are standing

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, MD, Principal Investigator — Department Of Otolaryngology
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be shared from university depository